CLINICAL TRIAL: NCT03724799
Title: The Investigation of Therapeutic Effect and Molecular Mechanism After Intravascular Laser Irradiation of Blood
Brief Title: Therapeutic Effect of Intravascular Laser Irradiation of Blood
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tri-Service General Hospital (Other)
Responsible Party: Principal Investigator, Cheng-Chiang Chang, Principal Investigator, Tri-Service General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: MOST 107-2314-B-016-074 -
Record Dates: First submitted 2018-10-28; First posted 2018-10-30 (Actual); Last update posted 2018-11-16 (Actual); Status verified 2018-11

CONDITIONS: Low-Level Laser Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- single arm (Experimental): Intravenous low level laser therapy
  Interventions: Device: Intravascular laser irradiation of blood for the patients with cerebral infarction

INTERVENTIONS:
Device: Intravascular laser irradiation of blood for the patients with cerebral infarction — Intravenous low level therapy has been a variety of applications in many different areas of medicine with a growing interest. It possesses laser specific biomodulation, analgesic, spasmolytic and even sedative effects among many other.

SUMMARY:
The investigators' previous studies results showed that the non-invasive treatment effects of low-energy lasers with the period of 5 consecutive days, could significantly improve the local function of static and dynamic motion stability of the lower extremities (p<0.0001) among the participants with lower limb periostitis. Therefore, investigators would like to further understand the treatment effect of intravascular low-energy laser on the central nervous system disorders. It is hoped that with this study, investigators can better understand how to use intravenous laser therapy to help those participants improve their ability of self-care and functional recovery.

ELIGIBILITY:
Healthy controls

Inclusion Criteria:

* Written informed consent that is consistent with ICH-GCP guidelines(The International Conference on Harmonisation's Guideline for Good Clinical Practice).
* Age ≥ 18 years and ≤80 years of age.
* Body weight ≥40 kg

Exclusion Criteria:

* Subjects with cranial metallic implants, cardiac pacemakers or claustrophobia.
* Previous diagnosis of stroke or dementia
* Significant history of depression
* History of symptomatic stroke
* History of seizures
* History or presence of any other major neurological disease
* Myocardial infarction within prior 6 months.
* Known presence of any malignancy
* Patients with bleeding tendency or coagulation profile abnormalities
* Have a serious infection or other serious medical illness that requires treatment and/or hospitalization within 90 days before study entry.
* Have received any of the following within 6 months of study entry: systemic corticosteroids; chemotherapy or radiation; erythropoietin, granulocyte colony-stimulating factor (G-CSF), granulocyte-macrophage colony-stimulating factor (GM-CSF), or growth hormone; drugs that affect the immune system including thalidomide, interleukins, interferons, or other cytokines; anabolic steroids at high levels; or any experimental agent, unless allowed otherwise by the researchers.
* Participation in any other investigational trial within 4 weeks of initial screening and within 7 weeks of study entry
* Contraindications to head CT, MRI, or SPECT
* Pregnant or lactating
* Botox treatment to the involved arm within three months of enrollment
* Subjects with conscious disturbance or moderate to severe aphasia

Stroke group:

Inclusion Criteria:

* Written informed consent that is consistent with ICH-GCP guidelines.
* Age ≥ 18 years and ≤80 years of age. Substantial unilateral motor impairment
* At least 6 months post thromboembolic ischemic stroke in subcortical region of MCA or lenticulostriate artery with or without cortical involvement.
* Between 6 and 24 months post-stroke, and having a motor or sensory neurological deficit
* No significant further improvement with physical therapy/rehabilitation
* Able and willing to undergo computed tomography (CT), magnetic resonance imaging (MRI), and single photon emission tomography (SPECT) scans of the head

Exclusion Criteria:

* History of more than 1 symptomatic stroke
* History of seizures
* History or presence of any other major neurological disease
* Myocardial infarction within prior 6 months.
* Known presence of any malignancy
* Patients with bleeding tendency or coagulation profile abnormalities
* Have a serious infection or other serious medical illness that requires treatment and/or hospitalization within 90 days before study entry.
* Have received any of the following within 6 months of study entry: systemic corticosteroids; chemotherapy or radiation; erythropoietin, granulocyte colony-stimulating factor (G-CSF), granulocyte-macrophage colony-stimulating factor (GM-CSF), or growth hormone; drugs that affect the immune system including thalidomide, interleukins, interferons, or other cytokines; anabolic steroids at high levels; or any experimental agent, unless allowed otherwise by the researchers.
* Participation in any other investigational trial within 4 weeks of initial screening and within 7 weeks of study entry
* Contraindications to head CT, MRI, or SPECT
* Pregnant or lactating
* Botox treatment to the involved arm within three months of enrollment
* Subjects with conscious disturbance or moderate to severe aphasia

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2018-11-14 (Estimated); Primary Completion 2019-09-30 (Estimated); Study Completion 2019-09-30 (Estimated)

PRIMARY OUTCOMES:
microcirculatory function of the skin | 12 days
  Laser Doppler Flowmetry is reliable for assessing microcirculatory status.

CONTACTS AND LOCATIONS:
Overall Officials: Cheng-Chiang Chang, MD. PhD., Principal Investigator — Tri-Service General Hospital

IPD SHARING:
Plan to Share IPD: No